CLINICAL TRIAL: NCT06286709
Title: FARGO: A Randomised, Phase IIa, Multi-centre, Placebo-controlled Trial of FAecal Microbiota Transplantation in primaRy sclerosinG chOlangitis
Brief Title: FAecal Microbiota Transplantation in primaRy sclerosinG chOlangitis
Acronym: FARGO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: PSC Support (Unknown); Life Arc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG_22-063
Record Dates: First submitted 2024-02-07; First posted 2024-02-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-05

CONDITIONS: Primary Sclerosing Cholangitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Cholangitis, Sclerosing; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Phase IIa, multi-centre, randomised, placebo-controlled, single-blinded, parallel group, clinical trial
Who Masked: Participant, Investigator
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Faecal Microbiota Transplant (FMT) (Active Comparator): FMT is 50mL aliquots of filtered suspension of stool (0.6g/mL). FMT for administration via colonoscopy will be made up of 150g stool in 250mL (5 aliquots). FMT for administration via enema will be made up of 30g stool in 50mL (1 aliquot) made up to 100mL by the addition of 50mL normal saline
  Interventions: Biological: Faecal Microbiota Transplant
- FMT Placebo (Placebo Comparator): FMT Placebo is 50mL aliquots of 0.9% w/v saline and glycerol in a ratio of 9 parts saline: 1 part glycerol v/v.
  Interventions: Other: FMT Placebo

INTERVENTIONS:
Biological: Faecal Microbiota Transplant — FMT is 50mL aliquots of filtered suspension of stool (0.6g/mL). FMT for administration via colonoscopy will be made up of 150g stool in 250mL (5 aliquots). FMT for administration via enema will be made up of 30g stool in 50mL (1 aliquot) made up to 100mL by the addition of 50mL normal saline
  Arms: Faecal Microbiota Transplant (FMT)
Other: FMT Placebo — FMT Placebo is 50mL aliquots containing 0.9% w/v saline and glycerol in a ratio of 9 parts saline: 1 part glycerol v/v. FMT Placebo for administration via colonoscopy will be made up of 250mL (5 aliquots). FMT Placebo for administration via enema will be made up of 50mL (1 aliquot) made up to 100mL by the addition of 50mL normal saline
  Arms: FMT Placebo

SUMMARY:
FARGO is a randomised, phase IIa, multi-centre, placebo-controlled trial to compare Faecal Microbiota Transplant (FMT) with placebo in patients with primary sclerosing cholangitis (PSC) and concomitant inflammatory bowel disease.

DETAILED DESCRIPTION:
Primary Sclerosing Cholangitis (PSC) is a chronic liver disease and there is no medical therapy proven to slow disease progression. Many patients with PSC also develop inflammatory bowel disease (IBD). It has been shown that there is an imbalance of 'normal' microbiome (e.g. bacteria, viruses, fungi) in the gut of people with PSC and IBD. This imbalance is believed to contribute to the development (and possibly worsening) of liver disease in PSC.

It is believed that Faecal Microbiota Transplant (FMT) treatment can restore the balance in the gut microbiome and that this can lead to reduction in symptoms of PSC and IBD and improve quality of life.

FMT involves the transplantation of faeces (or stool) from a healthy individual to a person with PSC. FMT is prepared from stool collected from unrelated, anonymous, healthy donors. The stool is treated in a laboratory at the University of Birmingham. The donors are carefully screened and the donated stool carefully tested to ensure that it is as clean and safe as possible before it is made into doses of FMT suitable for treatment purposes. Data from treatment with FMT in other conditions including Inflammatory Bowel Disease (IBD), Clostridioides difficile (C.diff) infection and PSC has shown FMT to be safe.

The primary aim of the FARGO trial is to determine the efficacy of FMT in patients with PSC. The FARGO trial will recruit 58 patients. Half will be randomised to FMT and half to placebo. The trial will be offered at a number of hospitals across England. Patients will be involved in the trial for 50 weeks, including a 2-week screening, 8 treatments over 8 weeks, and follow-up to 48 weeks post-randomisation. Trial visits will include the collection of health history, blood tests, stool tests, pregnancy tests (if applicable), medication reviews, disease specific measures, patient questionnaires and possible symptom and side-effect review. Research blood, urine, stool and colonic biopsy samples will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥ 18 years
3. Participants must be able to understand and comply with the purpose and procedures that are involved in the trial
4. An established diagnosis of colonic inflammatory bowel disease, with willingness to participate in an annual colonoscopic surveillance program, as per routine standard of care
5. An established clinical diagnosis of large duct PSC, with compatible features as assessed by magnetic resonance cholangiopancreatography (MRCP) or endoscopic retrograde cholangiopancreatography (ERCP)
6. A persistent ALP value above normal (at least 2 readings at this value over 6 months before screening)
7. Evidence of early to moderate stage liver fibrosis, as suspected by any of the following:

   1. Median VCTE score of ≤14.4kPa, with an interquartile range ≤30%
   2. Previous liver biopsy indicating at an absence of established cirrhosis, Ishak fibrosis stage <IV (or equivalent) in the last 24 months
   3. Serum enhanced liver fibrosis score (ELF) ≤9.8
8. A colonoscopy showing no evidence of dysplasia/neoplasia within 24 months before screening
9. No evidence of active colitis, as evidenced by a Partial Mayo Score of ≤4, with a score of <2 on the rectal bleeding domain at screening
10. Individuals with IBD who are receiving treatment with biologics, immunosuppression or corticosteroids must be taking a stable dose for at least twelve weeks prior to screening, and be expected to remain on the same medication/same dose for the duration of the trial
11. Individuals with PSC having overlapping features of autoimmune hepatitis may be included, provided:

    1. The dosage of immunosuppression has remained stable for at least twelve weeks prior to screening, and be expected to remain on the same medication/same dose for the duration of the trial; and
    2. There is evidence of concomitant colitis

Exclusion Criteria:

1. Secondary causes of sclerosing cholangitis including, but not limited to, IgG4-related cholangitis, cholangiopathy due to acquired immunodeficiency syndrome, drug-induced sclerosing cholangitis, trauma, ischaemic cholangiopathy, choledocholithiasis (investigator discretion), or sclerosing cholangiopathy as a sequelae of hepatopancreatobiliary resection
2. Other causes of liver disease, including, but not limited to, IgG4-related disease; viral hepatitis; alcohol-related liver disease; clinically significant metabolic associated fatty liver disease (at investigator discretion); drug-induced liver disease; hereditary haemochromatosis; alpha-1-antitrypsin disease; primary biliary cholangitis; Wilson disease; Budd-Chiari Syndrome; or primary or secondary hepatopancreatobiliary cancer
3. Presence of a clinically significant dominant stricture based on the combination of radiological, biochemical and clinical features. Patients can be included in the trial with a dominant extrahepatic stenosis if it has been stable for 6 months or more (as evidenced on imaging and also clinically), and one of the following are satisfied:

   1. The PI does not plan for any biliary intervention (endoscopic, percutaneous or surgical) for the duration of the trial OR
   2. The investigator decides that they do not wish to perform any biliary intervention (endoscopic, percutaneous or surgical) on the dominant stenosis for clinical reasons of stability/patient choice
4. Presence of a percutaneous drain or bile duct stent
5. Evidence of hepatic decompensation within twelve weeks prior to screening; or concern by the Principal Investigator that the participant may decompensate during the trial period. Hepatic decompensation as evidenced by variceal haemorrhage, ascites, hepatic hydrothorax, or hepatic encephalopathy (Appendix 1)
6. Biochemical/laboratory evidence of very advanced hepatic dysfunction, as evidenced by a serum bilirubin value >55 µmol/L (unless Gilbert Syndrome or another condition associated with unconjugated hyperbilirubinaemia, including but not limited to, spherocytosis and disorders of bilirubin conjugation where a bilirubin value>45 µmol/L is allowable), serum albumin <32 g/L, platelet level of <140x109/L, Child-Turcotte-Pugh (CTP) score >B7, or a MELD score >15
7. Ascending cholangitis as assessed clinically within twelve weeks of screening
8. Use of antibiotics within twelve weeks of screening
9. Participant already listed for liver transplantation, or concerns (investigator discretion) that they may need to be listed for liver transplantation during the trial period
10. Small duct PSC
11. Advanced-stage liver fibrosis, as evidenced by a VCTE score >14.4kPa, a liver biopsy showing >Ishak stage III fibrosis (or equivalent)
12. Significant renal dysfunction as evidenced by an estimated glomerular filtration rate of <60 ml/min according to the Cockcroft-Gault formula, or need for dialysis
13. Human Immunodeficiency Virus (HIV) infection
14. A symptomatic positive test result for Serious Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in the four weeks prior to screening
15. History of malignancy within the past three years, or ongoing malignancy, other than non-melanomatous skin cancer, or treated cervical carcinoma in situ
16. Any history of small bowel or colonic resection, or likelihood of resection during the trial period. Individuals with a sub-total colectomy and ileal pouch anal anastomosis are permitted to participate.
17. Patients who are pregnant or breastfeeding
18. Women of childbearing potential (see Appendix 2 for definition) who confirm they are not willing to practise effective contraception (see Appendix 3 for further details) for the duration of the trial and for four weeks after the last dose of trial drug. Women who are taking hormonal contraception must confirm stable formulation and dosage for at least 6 weeks prior to treatment
19. Alcohol consumption >21 units per week for men, and >14 units per week for women.
20. Positive urine drug screen at screening
21. Positive stool test for Clostridioides Difficile toxin or microscopy/culture positivity for enteric infection within twelve weeks prior to screening
22. Participation in an interventional trial, or use of a non-licensed investigational agent for any indication within twelve weeks before screening, or five half-lives of the investigational drug, whichever is longer
23. Newly introduced or a change in dosage of any of the following medications within twelve weeks of screening: fibric acid derivatives, farnesoid X-receptor agonists, anti-gastrointestinal motility agents (e.g., loperamide or opioids), bile acid sequestrants (e.g. colestyramine) or ursodeoxycholic acid (UDCA)
24. Use of any of the following medications within twelve weeks of screening: oral or intravenous antibiotics, including (but not limited to) vancomycin, rifaximin, rifampicin and metronidazole; probiotic or prebiotic preparations, including (but not limited to) VSL#3 and Symprove

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-29 (Estimated)

PRIMARY OUTCOMES:
Serum Alkaline Phosphatase (ALP) | ALP at Screening (Week -2), Week 1, Week 3, Week 5, Week 8, Week 12, Week 24, Week 36 and Week 48
  Reduction in serum ALP values from baseline, measured at 48 weeks following the first dose of FMT or FMT Placebo.

SECONDARY OUTCOMES:
Patient-reported outcome (PRO) measures | PSC-PRO at Screening (Week -2), Week 8, Week 12, Week 24, Week 36 and Week 48
  Patient-reported outcome (PRO) measure: Primary Sclerosing Cholangitis -Patient Reported Outcome (PSC-PRO) Questionnaire
Patient-reported outcome (PRO) measures | SF-36 at Screening (Week -2), Week 8, Week 12, Week 24, Week 36 and Week 48
  Patient-reported outcome (PRO) measure: short-form (SF)-36 Questionnaire
Patient-reported outcome (PRO) measures | 5D-Itch at Screening (Week -2), Week 8, Week 12, Week 24, Week 36 and Week 48
  Patient-reported outcome (PRO) measures: 5 dimensional itch scale (5D itch) Questionnaire
Patient-reported outcome (PRO) measures | SIBDQ at Screening (Week -2), Week 8, Week 12, Week 24, Week 36 and Week 48
  Patient-reported outcome (PRO) measures: Short Inflammatory Bowel Disease Questionnaire (SIBDQ)
Surrogate biomarkers of liver fibrosis | Surrogate biomarkers of liver fibrosis: VCTE at Screening (Week -2) and Week 48
  Surrogate biomarkers of liver fibrosis: vibration-controlled transient elastography (VCTE)
Surrogate biomarkers of liver fibrosis | Surrogate biomarkers of liver fibrosis: ELF at Week 1, Week 5, Week 12, and Week 48
  Surrogate biomarkers of liver fibrosis: enhanced liver fibrosis score (ELF)
Routine liver laboratory parameters | Routine liver laboratory parameters: ALT at Screening (Week -2), Week 1, Week 3, Week 5, Week 8, Week 12, Week 24, Week 36 and Week 48
  Routine liver laboratory parameters: serum alanine transaminase (ALT)
Routine liver laboratory parameters | Routine liver laboratory parameters: AST at Screening (Week -2), Week 1, Week 3, Week 5, Week 8, Week 12, Week 24, Week 36 and Week 48
  Routine liver laboratory parameters: serum aspartate aminotransferase (AST)
Routine liver laboratory parameters | Routine liver laboratory parameters: bilirubin at Screening (Week -2), Week 1, Week 3, Week 5, Week 8, Week 12, Week 24, Week 36 and Week 48
  Routine liver laboratory parameters: bilirubin
Routine liver laboratory parameters | Routine liver laboratory parameters: gamma glutamyl transferase at Screening (Week -2), Week 1, Week 3, Week 5, Week 8, Week 12, Week 24, Week 36 and Week 48
  Routine liver laboratory parameters: gamma glutamyl transferase
Routine liver laboratory parameters | Routine liver laboratory parameters: albumin at Screening (Week -2), Week 1, Week 3, Week 5, Week 8, Week 12, Week 24, Week 36 and Week 48
  Routine liver laboratory parameters: albumin
PSC specific prognostic scores | PSC specific prognostic scores: UK-PSC Score at Screening (Week -2), Week 1, Week 3, Week 5, Week 8, Week 12, Week 24, Week 36 and Week 48
  PSC specific prognostic scores: the UK-PSC Score
PSC specific prognostic scores | PSC specific prognostic scores: Amsterdam-Oxford PSC Score at Screening (Week -2), Week 1, Week 3, Week 5, Week 8, Week 12, Week 24, Week 36 and Week 48
  PSC specific prognostic scores: the Amsterdam-Oxford PSC score
Quantitative assessment of Inflammatory Bowel Disease (IBD) activity | Quantitative assessment of IBD activity: Mayo colitis score at Week 1, Week 12 and Week 48
  Quantitative assessment of IBD activity: The Mayo colitis score
Quantitative assessment of IBD activity | Quantitative assessment of IBD activity: SES-CD at Week 1, Week 12 and Week 48
  Quantitative assessment of IBD activity: The Simple Endoscopic Score for Crohn's Disease (SES-CD);
Quantitative assessment of IBD activity | Quantitative assessment of IBD activity: faecal calprotectin at Screening (Week -2), Week 1, Week 5, Week 12 and Week 48
  Quantitative assessment of IBD activity: faecal calprotectin
The incidence of clinical non-trial endpoint events | The incidence of clinical non-trial endpoint events at Screening (Week -2), Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 12, Week 24, Week 36 and Week 48
  The incidence of clinical non-trial endpoint events: acute cholangitis flares (including those that are resistant to single course antibiotic treatment), acute colitis flares, and episodes/time to hepatic decompensation
The incidence of trial endpoint events | The incidence of trial endpoint events at Screening (Week -2), Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 12, Week 24, Week 36 and Week 48
  The incidence of trial endpoint events: cholangiocarcinoma / hepatopancreatobiliary malignancy, referral for liver transplantation, colonic resection or colorectal cancer, and/or mortality
Occurrence of adverse events | Occurrence of adverse events at Screening (Week -2), Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 12, Week 24, Week 36 and Week 48
  Occurrence of adverse events as measured by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - St Mark's Hospital, London North West University Healthcare NHS Trust, London
  - Royal Free Hospital, Royal Free London NHS Foundation Trust, London
  - King's College Hospital, King's College Hospital NHS Foundation Trust, London
  - John Radcliffe Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient level data may be shared in accordance with the Cancer Research UK Clinical Trials Unit (CRCTU) Data Sharing Policy. More detailed information on the CRCTU's Data Sharing Policy and the mechanism for obtaining data can be found on the CRCTU website:
  https://www.birmingham.ac.uk/research/crctu/data-sharing-policy
Supporting Information: Study Protocol
URL: https://www.birmingham.ac.uk/research/crctu/data-sharing-policy

REFERENCES:
- [Derived] Al-Shakhshir S, Quraishi MN, Mullish B, Patel A, Vince A, Rowe A, Homer V, Jackson N, Gyimah D, Shabir S, Manzoor S, Cooney R, Alrubaiy L, Quince C, van Schaik W, Hares M, Beggs AD, Efstathiou E, Rimmer P, Weston C, Iqbal T, Trivedi PJ. FAecal micRobiota transplantation in primary sclerosinG chOlangitis (FARGO): study protocol for a randomised, multicentre, phase IIa, placebo-controlled trial. BMJ Open. 2025 Jan 6;15(1):e095392. doi: 10.1136/bmjopen-2024-095392. PMID 39762111